CLINICAL TRIAL: NCT05446649
Title: Dry Needling Versus Instrumented Assisted Soft Tissue Mobilization In the Patient With Cervicogenic Treatment Headache; Randomized Controlled Trial
Brief Title: Dry Needling Versus Instrumented Assisted Soft Tissue Mobilization In the Patient With Cervicogenic Treatment Headache
Acronym: DN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Al Shaymaa Shaaban Abd El Azeim, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: p.t.rec/012/003725
Record Dates: First submitted 2022-06-26; First posted 2022-07-07 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cervicogenic Headache
Keywords: dry needling; cervicogenic headache; instrumented assisted soft tissue mobilization
MeSH Terms: conditions — Post-Traumatic Headache | interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: dry needling and instrumented assisted soft tissue mobilization
Who Masked: Participant, Outcomes Assessor
Masking Description: random generator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- dry needling (Experimental): the patient will receive dry needling and conventional therapy three times per week for four weeks
  Interventions: Other: dry needling; Other: conventional therapy
- instrumented assisted soft tissue mobilization (Experimental): the patient will receive instrumented assisted soft tissue mobilization and conventional therapy three times per week for four weeks
  Interventions: Other: instrumented assisted soft tissue mobilization; Other: conventional therapy
- conventional therapy (Active Comparator): the patient will receive conventional therapy three times per week for four weeks
  Interventions: Other: conventional therapy

INTERVENTIONS:
Other: dry needling — the patient will be in comfortable position .and clean the area over upper trapezius and sub occipital muscles. detect the trigger point then Perpendicular needling into the bulk of the muscle is the safest technique for this area.
  Arms: dry needling
Other: instrumented assisted soft tissue mobilization — the patients will be in sitting position. The appropriate IASTM technique instrument will be selected to scan, and then treat the affected area for 30 to 60 seconds per treated area. The procedure will be applied to the superficial cervical fascia and investing the layers of deep cervical fascia that surround all the structures in the neck. Strokes will be applied on the sub occipital and upper fibers of trapezius muscle. The IASTM technique will be applied at a 45° angle in a direction parallel to the treated muscle fibers for 20 seconds, followed immediately by an additional 20 seconds application at a 45° angle in a perpendicular direction to the muscle fibers, resulting in a total treatment time of approximately 40 seconds. The patients will be advised that they might be sore, bruised, or have small red dots called petechiae, on the treated area. Ice will be applied for 15 to 20 min after the treatment if there will be a massive soreness.
  Arms: instrumented assisted soft tissue mobilization
Other: conventional therapy — patients will be received traditional physiotherapy (stretching and strengthening cervical muscles and postural correction exercise)

SUMMARY:
the aim of this study is to investigate the efficacy of Dry Needling Versus Instrumented Assisted Soft Tissue Mobilization In the Patient With Cervicogenic Treatment Headache

DETAILED DESCRIPTION:
Cervicogenic headache has been classified as a secondary type headache, and it is usually associated with cervical myofascial pain sources as myofascial trigger points . It also could be related to any joint, disc, and ligament disease of the upper region of the neck.physiotherapist use trigger point dry needling as an invasive treatment for CGH where a solid filament needle is inserted into a myofascial trigger point . The advantages of Dry needling are increasingly documented .Instrument-assisted soft tissue mobilization technique has been reported to decrease pain, improve overall function, and increase range of motion . It enhances the ability of physical therapists to detect altered tissue properties, through the vibration sense within the instrument, and to treat soft tissue dysfunction. It also enhances the patient's awareness of altered sensations within the treated tissues.

ELIGIBILITY:
Inclusion Criteria:

* 20 to 60 years old patient with unilaterally of the head pain
* pain triggered by external pressure over the upper cervical joints (c1-c3)
* pain elicited by the neck movements, and/or sustained awkward positions with reduced neck ROM
* headache intensity pain score of at least 20mm on the Visual analogue scale (VAS)
* headache frequency of at least once a week for at least 3 months
* minimum neck disability index score of 10 points or greater

Exclusion Criteria:

* Migraine, tension- type headache, tumor, osteoporosis, fracture, rheumatoid arthritis and metabolic diseases.
* Prolonged history of steroid use.
* Resting blood pressure greater than 140/90 mmhg.
* cervical spinal stenosis, diminished sensation and central nervous system involvement,
* previous head or neck surgery or whiplash injury history within the last 6 weeks

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-08-30 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
pain intensity | up to four weeks
  visual analogue scale will be used to asses pain intensity which patient will be instructed to put point on line from no pain to tolerable pain. The scale consists of a line, usually 10 cm long, ranging from no pain or discomfort (zero) , to the worst pain that could possibly feel .
neck disability | up to four weeks
  will be measured by Arabic neck disability index. It contains ten category/classes. Each category contains six choices (zero-five).Score from zero to four no disability, from five to 15 this is mild, From 15 to 24 this is moderate, from 25 to 34 this is severe, more than 34 this is a complete disability
pressure pain threshold | up to four weeks
  pressure pain threshold will be assessed by commander algometer

SECONDARY OUTCOMES:
range of motion | up to four weeks
  range of motion will be measured by inclinometer CROM. The CROM (deluxe version - Performance Attainment Associates, Roseville, MN, USA) measures the cervical range of motion5- for ﬂexion, extension, lateral ﬂexion, and rotation using separate inclinometers. These inclinometers are attached to a frame similar to that for eyeglasses one in the sagittal plane for ﬂexion - extension, second in the frontal plane for lateral ﬂexion and a third in the horizontal plane for rotation.
headache frequency | up to four weeks
  the number of days the subjects feel headache (headache frequency).
medication intake | up to four weeks
  from the patients' diary in the last week , medications intake will be recorded as follow: 1) not at all; 2) once a week; 3) once every couple of days; 4) once or twice a day; or 5) three or more times a day
headache duration | up to four weeks
  the total hours of headache (headache duration).

CONTACTS AND LOCATIONS:
Locations (1):
- Alshaymaa Shaaban Abd El-Azeim, Giza, Egypt

REFERENCES:
- [Derived] Elhafez HM, Mohammed OA, Fahmy EM, Elkhateeb YS, Abd El-Azeim AS. Dry needling versus instrument assisted soft tissue mobilization in patients with cervicogenic headache: a randomized controlled trial. Disabil Rehabil. 2025 Dec 23:1-13. doi: 10.1080/09638288.2025.2605621. Online ahead of print. PMID 41437643